CLINICAL TRIAL: NCT03072056
Title: A Phase 1, Open-Label, 3-Period, Single-Ascending Dose, Crossover Study in Healthy Subjects to Compare PK Properties of MIN-101 and Its Metabolites Poor and Extensive Metabolizers as Defined by Cytochrome P450 2D6 Genotype
Brief Title: A Pharmacokinetic Study of MIN-101 and Its Metabolites in Healthy Subjects to Compare MIN-101 in Poor and Extensive Metabolizers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Minerva Neurosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MIN-101C05
Record Dates: First submitted 2017-02-23; First posted 2017-03-07 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — roluperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Extensive Metabolizers, 4 mg (Experimental): subjects will receive 32 mL of MIN-101 as a 0.125 mg/mL oral solution
  Interventions: Drug: MIN-101
- Extensive Metabolizers, 8 mg (Experimental): subjects will receive 32 mL of MIN-101 as a 0.25 mg/mL oral solution
  Interventions: Drug: MIN-101
- Extensive Metabolizers, 16 mg (Experimental): subjects will receive 32 mL of MIN-101 as a 0.5 mg/mL oral solution
  Interventions: Drug: MIN-101
- Poor Metabolizers, 4 mg (Experimental): subjects will receive 32 mL of MIN-101 as a 0.125 mg/mL oral solution
  Interventions: Drug: MIN-101
- Poor Metabolizers, 8 mg (Experimental): subjects will receive 32 mL of MIN-101 as a 0.25 mg/mL oral solution
  Interventions: Drug: MIN-101
- Poor Metabolizers, 16 mg (Experimental): subjects will receive 32 mL of MIN-101 as a 0.5 mg/mL oral solution
  Interventions: Drug: MIN-101

INTERVENTIONS:
Drug: MIN-101

SUMMARY:
* To evaluate the pharmacokinetic (PK) profile of MIN-101 and its metabolites in extensive (EM) and poor (PM) metabolizers
* To evaluate the relationship between plasma levels of MIN-101 and changes in QT/QTcF intervals
* To evaluate safety and tolerability of MIN-101.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed CYP2D6 extensive or poor metabolizer genotype
2. Subject has given voluntary written informed consent before performance of any study related procedure
3. Subject must be 18 to 45 years of age, inclusive
4. Subject must be a healthy male or female as indicated by the following:

   * Clinical chemistries, hematology, and urinalysis tests must be within normal, allowable limits (if out of range, and with the exception of potassium, magnesium, and calcium, must be considered clinically significant to be exclusionary) and performed within 21 days of receiving first dose of study drug
   * Body mass index of between 18 and 30 kg/m2
   * Normal vital signs after 5 minutes resting in supine position and in standing position after 5 minutes of resting in supine position:

     * 95 mm Hg < systolic blood pressure < 140 mm Hg
     * 50 mm Hg < diastolic blood pressure < 90 mm Hg
     * 50 bpm < heart rate < 90 bpm
     * Systolic blood pressure decrease of less than 20 mm Hg within 3 minutes of standing
     * Diastolic blood pressure decrease of less than 10 mm Hg within 3 minutes of standing
   * Normal 12-lead automatic ECG: 120 ms < PR < 210 ms, QRS < 120 ms, QTc (Fridericia) ≤ 430 msec for males and ≤ 440 ms for females
5. Agree to abstain from all medication (except for allowed birth control in #5 below), including non-prescription and prescription medication (including vitamins and natural or herbal remedies, e.g. St. John's Wort) for 21 days before the first study day until discharge from the study (end of post study medical).
6. Subject agrees to use an adequate method of birth control (excluding oral hormonal contraception). Subjects who are sexually active must use, with their partner, 2 approved methods of highly effective contraception from the time of study drug administration until 90 days after the last dose of study drug.

Exclusion Criteria:

1. A history of clinically significant gastrointestinal disease, especially peptic ulcerations, gastrointestinal bleeding, ulcerative colitis, Crohn's disease or Irritable Bowel Syndrome; renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic or psychiatric disease, especially those with a past history of depression, suicidal ideation or suicide attempts, or cardiovascular disease, or any other condition which, in the opinion of the principle investigator, would jeopardize the safety of the subject or impact the validity of the study results
2. Acute diarrhea or constipation in the 7 days before the predicted first study day. If screen occurs > 7 days before first study day, this criterion will be determined on first study day.
3. Subject has donated blood within 90 days or plasma within 30 days of study dosing
4. Regular alcohol consumption in males > 21 units per week and females > 14 units per week (1 Unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
5. Subject has a borderline or long QTc interval by the Fridericia correction method, as defined by screening readings of > 430 msec for males and > 440 for females or a personal or familial history of long QT syndrome
6. Subject has participated in a clinical trial within 90 days prior to study initiation
7. Females of child bearing potential who are pregnant, breast feeding or who are either not surgically sterile, postmenopausal, or are sexually active and not using an acceptable form of contraception
8. Subject has used any over-the-counter (OTC) medication, dietary or herbal supplements, including vitamins, within 21 days prior to study entry
9. Subject has used any prescription medication within 21 days prior to the Day -1
10. Subject has been treated with any known CYP2D6 or CYP3A4 enzymes altering drugs within 30 days prior to the study
11. Subject has smoked or used tobacco products within 2 months prior to or during the study
12. Subject has sought advice from or been referred to a GP or counselor for abuse or misuse of alcohol, non-medical drugs, medicinal drugs or other substance abuse, e.g.

    solvents
13. Subject has a positive blood screen for HIV, Hepatitis B surface antigen (HBsAg), and Hepatitis C antibody and/or a positive urine screen for drugs of abuse or positive alcohol breath test at screening, or history of positive urine drugs of abuse screens
14. Any current or previous use of drugs such as opiates, cocaine, ecstasy, or intravenous amphetamines Subjects who admit to occasional past use of cannabis will not be excluded as long as they have a negative drugs-of-abuse test and have been abstinent from cannabis use for at least 3 months
15. Subject has an uncontrolled inter-current illness (i.e., active infection)
16. Subject has had major surgery within 28 days of study entry, or 12 months prior to study for gastrointestinal surgery.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Plasma PK parameter, Cmax | 0, .25, .5, .75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 14, 16, 24, 28, 32, 36, 48, 52, 56, 60, 72, and 76 hr post-dose on Day 1 of 3 periods (each period is up to 6 days). One sample from PM subjects at hr 98±2
  To estimate the relative bioavailability of MIN-l0l following MIN-101 administration. Plasma samples will be analyzed for MIN-101 and its metabolites using a validated LC-MS/MS method
Plasma PK parameter, Tmax | from predose up to 76 hours post dose
Plasma PK parameter, Tlag | from predose up to 72 hours post dose
Plasma PK parameter,partial AUC (e.g., AUC12, AUC24), AUClast, AUC∞ | from predose up to 72 hours post dose
Plasma PK parameter, λz and t1/2 | from predose up to 72 hours post dose
To evaluate the relationship between plasma levels of MIN-101 and its main metabolites and changes in QT/QTcF intervals in healthy CYP2D6 EM and PM subjects | at -1.5, -1, -0.25 (predose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 28, 32, 36, 48, 56, 72, and 76 hours post-dose on Day 1 of the 3 periods (each period is up to 6 days).

SECONDARY OUTCOMES:
Safety (AE reporting, safety laboratory parameters analysis, vital signs and 12 lead ECG assessments) | 3 months and 7 days
  Safety will be assessed through AE reporting, safety laboratory parameters analysis, vital signs and 12 lead ECG assessments

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jabbari, MD, Principal Investigator — BioKinetic Europe Ltd
Locations (1):
- Biokinetic Europe, Belfast, Ireland

IPD SHARING:
Plan to Share IPD: No